CLINICAL TRIAL: NCT06131684
Title: Utility of Amniotic Fluid Analysis for Intrapartum Infection Prediction Model
Brief Title: Amniotic Fluid Analysis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Croslanda, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00024844
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrauterine pressure catheter (IUPC) present (Active Comparator): An IUPC is placed through the standard of care.
  Interventions: Device: Intrauterine pressure catheter (IUPC) present
- Intrauterine pressure catheter (IUPC) absent (Active Comparator): No IUPC is required
  Interventions: Device: Intrauterine pressure catheter (IUPC) absent

INTERVENTIONS:
Device: Intrauterine pressure catheter (IUPC) present — Amniotic fluid will be analyzed every 3 hours for the duration of labor for patients who require an IUPC through the standard of care.
  Arms: Intrauterine pressure catheter (IUPC) present
Device: Intrauterine pressure catheter (IUPC) absent — Patients that do not require an IUPC through the standard of care will not have amniotic fluid analyzed.
  Arms: Intrauterine pressure catheter (IUPC) absent

SUMMARY:
This is a prospective study that will aid in ensuring the feasibility of timely and correct aspiration of amniotic fluid by study research team that include the clinical team taking care of the patient during her labor, timely transport and interpretation of specimens. It will also assist in providing information for the computation of necessary statistical measures (e.g. sample size, power analysis, etc.) for the study cohorts that lack the needed data in the medical literature.

DETAILED DESCRIPTION:
Can amniotic fluid be serially aspirated via an Intrauterine pressure catheter (IUPC) and successfully analyzed in labor? Do abnormal amniotic fluid results collected serially predict which laboring patients will develop an intrapartum infection? Can the results predict infection sooner than the current clinical diagnostic criteria as outlined by the 2015 NICHD guidelines? How do the sensitivity, specificity, positive and negative predictive values compare to the 2015 NICHD diagnostic criteria?

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age ≥ 37 weeks
* Age of participant ≥ 18 years old

Exclusion Criteria:

* Multiple gestation
* Gestational age < 37 weeks
* Intrauterine fetal demise
* Fetal anomalies
* Pre-gestational Diabetics / Gestational Diabetics
* Chronic immune suppression with steroids (defined as > 1 month of consistent steroid use)
* Oligohydramnios
* Women with documented non-obstetric infections within 2 weeks of admission; including use of any antibiotics within 2 weeks of admission for non-documented/suspected infections
* Repeat temperature not performed within 45 minutes of index fever (100.4 F)
* Index fever (100.4 F) is > 1 hour after delivery
* Expectantly managed premature rupture of membranes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients who develop an intrapartum infection | From enrollment to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Adam Crosland, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science Univerity, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No